CLINICAL TRIAL: NCT02227264
Title: Primary Hyperparathyroidism: Short-term Calcimimetics Treatment - Relevance for Parathyroid Surgery Decisions?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Inga-Lena Nilsson, M.D., Ph.D; Assoc.prof., Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2012-005374-57
Record Dates: First submitted 2014-08-17; First posted 2014-08-28 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Primary Hyperparathyroidism
Keywords: Primary hyperparathyroidism; Calcimimetic Agents; Parathyroid adenomectomy
MeSH Terms: conditions — Hyperparathyroidism, Primary | interventions — Cinacalcet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cinacalcet (Experimental): Cinacalcet, Mimpara®: 30 mgx1 for four weeks. In case of persistent hypercalcemia after two weeks of treatment with Mimpara® 30 mgx1, the dosage of Mimpara® will be increased to 60 mg daily.
  Second intervention: Parathyroid adenomectomy.
  Interventions: Drug: Cinacalcet; Procedure: parathyroid adenomectomy

INTERVENTIONS:
Drug: Cinacalcet — Cinacalcet, Mimpara® 30mgx1-2 for 4 weeks
  Other Names: H05BX01; Mimpara®
Procedure: parathyroid adenomectomy — surgical removal of pathologic parathyroid tissue

SUMMARY:
Patients with primary hyperparathyroidism (pHPT) often present with fatigue, psychological and cognitive symptoms. Improvement in these symptoms after parathyroid adenomectomy (PTX) has been reported. But physicians lack a method to attribute the symptoms to pHPT and to predict the reversibility after PTX.

This study aims to evaluate short-term calcimimetic treatment as a tool for predicting the outcome of PTX on muscle strength, quality of life, psychological symptoms, and cognitive function in patients with pHPT.

Material and Methods: 118 patients scheduled for PTX at Karolinska University Hospital, Sweden, will have a four week treatment with calcimimetics (Mimpara®) before undergoing surgery. Biochemicals, muscle strength, quality of life, psychological symptoms and cognitive function will be analysed at baseline, after four week follow-up and postoperatively.

Hypothesis: The outcome of short-term calcimimetic treatment can predict the outcome of PTX on muscle strength, quality of life, psychological symptoms, and cognitive function in patients with pHPT

DETAILED DESCRIPTION:
The study evaluates if short-term treatment with calcimimetics may be used for patients with PHPT as a relevant guide in the decision of when to choose parathyroid surgery, by predicting the outcome of surgical treatment.

120 ± 2 patients with primary hyperparathyroidism scheduled for parathyroid surgery will be included in the study after informed consent and will receive study medication with cinacalcet, Mimpara® 30 mgx1 for four weeks. In case of persistent hypercalcemia after two weeks of treatment with Mimpara® 30 mgx1, the dosage of Mimpara® will be increased to 60 mg daily. During the study drug treatment period, the patients will be followed closely at least once a week with clinical monitoring and control of serum ionized calcium, given the risk of side effects and hypocalcemia. If the concentration of ionized calcium in serum will decrease to a subnormal level (<1.15 mmol/l), the Mimpara® treatment will be discontinued temporarily and only reinserted in a lower dose (30 mg x 1) if the concentration of ionized calcium raises over 1.33 mmol/l. The size of the cohort has been decided after power estimations based on the results in study part A. Both groups will go through the test panel of self-rating scales described above at four occasions (Figure).

The Outcome to be registered are the changes from baseline to the end of the study medication period compared to the changes postoperatively, thus the changes between the Visit 2 to Visit 6 and the changes between Visit 2 and Visit 7 and Visit 8 respektively.

Assessments and Procedures Visit 1: Clinical examination (general condition, neck, blood pressure, cor et pulm). Screening of patients with primary hyperparathyroidism scheduled for parathyroid surgery. Patient that fulfills inclusion and exclusion criteria will be asked to participate in the study.

Visit 2: Informed consent is signed. Test panel of self rating scales (Quality of Life Questionnaire-Core 30 (QLQ-C30), Positive States of Mind (PSOM )and Hospital Anxiety and Depression scale (HAD), cognitive test (Montreal cognitive assessment (MoCA-Test)) and muscle strength (Timed stand test). Blood samples are drawn within 2 weeks before and analyzed for: parathyroid hormone (p-PTH), s-ionized calcium, p-total calcium, p-albumin, p-creatinine, p-phosphate, s-25-OH-D-vitamin and p-TSH. Initiation of treatment with Mimpara® 30 mg x 1. Clinical examination (general condition, blood pressure). For fertile women, a pregnancy test is demanded before enrollment.

Visit 3: Week 1 (± 2 days); blood samples for analysis of ionized calcium. History of symptoms related to hypocalcemia (paresthesias, cramps, muscle fatigue). Clinical examination when indicated (general condition, blood pressure).

Visit 4: Week 2 (± 2 days); blood samples for analysis of ionized calcium. History as above. Mimpara® continued, If the ionized calcium level is >1.33 mmol/l: increase of dosage of Mimpara® to 30 mg x 2.

Visit 5: Week 3 (± 2 days); blood samples for analysis of ionized calcium. History as above. Mimpara® treatment completed.

Visit 6 (3): Week 4 (± 2 weeks in study B); Test panel of self rating scales (QLQ-C30, PSOM and HAD), cognitive test (MoCA-Test) and muscle strength (Timed stand test). Blood samples are drawn and analyzed for: plasma (p)-PTH, serum(s)-ionized serum calcium, p-total calcium, p-albumin, p-creatinine, p-phosphate.

Visit 7 (4): Postoperative follow up, 6 (± 1 week) post surgery; Test panel of self rating scales (QLQ-C30, PSOM and HAD), cognitive test (MoCA-Test) and muscle strength (Timed stand test). Blood samples are drawn and analyzed for plasma p-PTH, s-ionized calcium, p-total calcium, p-albumin, p-creatinine, p-phosphate, s-25-OH-D-vitamin and p-TSH.

Visit 8 (5): Postoperatively, 6 months post surgery (± 3 weeks); Test panel of self rating scales (QLQ-C30, PSOM and HAD), cognitive test (MoCA-Test) and muscle strength (Timed stand test). Blood samples are drawn and analyzed for plasma (p)-PTH, s-ionized calcium, p-total calcium, p-albumin, p-creatinine, p-phosphate, s-25-OH-D-vitamin and p-TSH.

ELIGIBILITY:
Inclusion Criteria:

* Primary hyperparathyroidism
* Scheduled for parathyroid surgery
* Age >40
* Ability to participate in all tests included in the study model
* Signed consent

Exclusion Criteria:

* Pregnancy
* Breast feeding
* Fertile woman not using contraceptives (IUD or pills)
* Impaired kidney function, GFR < 40 ml/min
* Intolerance to Mimpara®
* Previously treated with Mimpara®
* Participating in other ongoing clinical study
* Epilepsy
* Severe hepatic impairment
* Hypotension
* Heart failure (NYHA class 3-4, symptoms with minimal exertion)
* Medication with ketoconazole (oral) or tricyclic antidepressants

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-06; Primary Completion 2021-12 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Predictive outcome in Quality of Life after parathyroidectomy | after four weeks of calcimimetic treatment and postoperatively
  Health related quality of life measured by EORTC QLQ-C30 (total score)

SECONDARY OUTCOMES:
Psychological well-being | After four weeks of calcimimetic treatment and postoperatively
  Psychological well-being, evaluated with the validated form Positive States of Mind, PSOM
Anxiety and depression | After four weeks of calcimimetic treatment and postoperatively
  Depression and anxiety; evaluated with the Hospital Anxiety and Depression (HAD) scale
Muscle strength | After four weeks of calcimimetic treatment and postoperatively
  Leg muscle strength measured by Timed stand-test (repeated uprise from chair)
Biochemical data | After four weeks of calcimimetic treatment and postoperatively
  AE/SAE recording and safety blood samples; serum levels of p-PTH, s-ionized calcium, p-total calcium, p-albumin, p-creatinine, p-phosphate, s-25-OH-D and thyroid-stimulating hormone (TSH)
Cognitive function | after four weeks of calcimimetic treatment and postoperatively
  Cognitive function evaluated with Montreal cognitive assessment (MoCA-test)

CONTACTS AND LOCATIONS:
Overall Officials: Inga-Lena Nilsson, M.D., Ph.D, Principal Investigator — Karolinska UH; Inga-Lena Y Nilsson, MD, PhD, Principal Investigator — Karolinska UH
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koman A, Ohlsson S, Branstrom R, Pernow Y, Branstrom R, Nilsson IL. Short-term medical treatment of hypercalcaemia in primary hyperparathyroidism predicts symptomatic response after parathyroidectomy. Br J Surg. 2019 Dec;106(13):1810-1818. doi: 10.1002/bjs.11319. Epub 2019 Oct 9. PMID 31595982
- See also: Karolinska University Hospital — http://www.karolinska.se/
- See also: Karolinska Institute — http://ki.se/
- See also: Ethical Review Board — http://www.epn.se